CLINICAL TRIAL: NCT06884540
Title: Optimizing Patient-centred Outcomes Using Opioid Minimization Strategies (OPUS) Anesthesia: a Pilot Randomised Controlled Trial
Brief Title: Optimizing Patient-centred Outcomes Using Opioid Minimization Strategies: The OPUS Anesthesia Pilot Trial
Acronym: OPUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Perioperative Anesthesia Clinical Trials (PACT) Group (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); International Anesthesia Research Society (IARS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMS-162
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia; Anesthesia Complication; Surgery; Quality of Life; Pain, Postoperative; Anesthesia Morbidity; Feasibility Studies; Patient-centredness
Keywords: Pilot trial; Anesthesia; Quality of recovery; Postoperative pain; Opioid minimization strategies; Dexmedetomidine; Lidocaine; Patient-centred outcomes
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Lidocaine; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intraoperative intravenous dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Intraoperative intravenous lidocaine (Experimental)
  Interventions: Drug: lidocaine
- Usual care (Other)
  Interventions: Other: control group

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous bolus: between 0.2 and 0.5 mcg/kg.
  followed by
  Intravenous infusion: ranging from 0.2 to 0.7 mcg/kg/h to the discretion of the attending anesthesiologist.
  Bolus will be initiated prior to surgical incision and infusion will be stopped at wound closure.
  Arms: Intraoperative intravenous dexmedetomidine
Drug: lidocaine — Intravenous bolus: between 0.5 and 1.5 mg/kg.
  followed by
  Intravenous infusion: ranging from 0.5 to 2.0 mg/kg/h to the discretion of the attending anesthesiologist.
  Bolus will be initiated prior to surgical incision and infusion will be stopped at wound closure.
  Arms: Intraoperative intravenous lidocaine
Other: control group — Usual care where systemic dexmedetomidine is not allowed and systemic lidocaine is permitted only for the prevention or treatment of propofol injection pain.
  Arms: Usual care

SUMMARY:
Up to 40% of patients experience suboptimal recovery in the days following major surgery, limiting their return to functional independence. Few preventive interventions exist, but intravenous dexmedetomidine and lidocaine administered during general anesthesia represent simple strategies that may significantly impact recovery and other patient-centred outcomes after surgery. The goal of this pilot trial is to determine the feasibility of conducting a phase 3 pragmatic adaptive multicentre trial to evaluate the impact of dexmedetomidine and lidocaine administered during major non-cardiac surgery on patient-centred outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults >/= 18 years.
2. Having elective major non-cardiac surgery (i.e., planned duration >/= 1.5 hours and anticipated >/= 1 night hospital stay).
3. Requiring general anesthesia.
4. Able to complete baseline quality of recovery assessment.

Exclusion Criteria:

1. Individuals with known contraindications to dexmedetomidine or lidocaine (e.g., allergy to alpha-2 agonists or local anesthetics, severe renal or hepatic failure, bradycardia or hypotension), as per routine assessment.
2. Regular use of alpha-2 agonists or local anesthetics prior to hospitalization.
3. Pregnant women.
4. Planned use of regional analgesia (i.e., epidural, peripheral nerve block, trunk nerve block) in conjunction with general anesthesia. Local anesthetics such as lidocaine are administered as part of regional analgesia technique. Combination with intravenous lidocaine is contraindicated to avoid exceeding therapeutic concentration.
5. Planned postoperative intubation after PACU discharge.
6. No fixed address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 week
  Number of patients who are approached to participate by the study team and who consent to participate in the study.

SECONDARY OUTCOMES:
Proportion of participants receiving dexmedetomidine | 24 hours
  Proportion of patients in the dexmedetomidine group who receive per protocol treatment (i.e. they receive dexmedetomidine during general anesthesia).
Proportion of participants receiving lidocaine | 24 hours
  Proportion of patients in the lidocaine group who receive per protocol treatment (i.e. they receive lidocaine during general anesthesia).
Completeness of data collection for outcome measures | 6 months
  Completeness of data collection, defined as the percentage of instruments or data fields completed with at least 90% of expected forms or relevant fields completed at each time point for each instrument and participant.
Sex representativeness of participants | 6 months
  Proportion of female participants enrolled in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Verret, MD PhD FRCPC, Principal Investigator — CHU de Quebec-Université Laval Research Center; Dean A. Fergusson, PhD, Principal Investigator — Ottawa Hospital Research Institute; Manoj M. Lalu, MD PhD FRCPC, Principal Investigator — Ottawa Hospital Research Institute; Alexis Turgeon, MD MSc FRCPC, Principal Investigator — CHU de Quebec-Université Laval Research Center
Locations (1):
- CHU de Québec-Université Laval (Hôpital de l'Enfant-Jésus), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No